CLINICAL TRIAL: NCT04434040
Title: A Single Arm Phase 2 Trial of Atezolizumab With Sacituzumab Govitecan to Prevent Recurrence in Triple Negative Breast Cancer (ASPRIA)
Brief Title: Atezolizumab + Sacituzumab Govitecan to Prevent Recurrence in TNBC (ASPRIA)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Genentech, Inc. (Industry); Stand Up To Cancer (Other)
Responsible Party: Principal Investigator, Elizabeth A Mittendorf, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-028
Record Dates: First submitted 2020-06-14; First posted 2020-06-16 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer; Triple Negative Breast Cancer; Residual Cancer; Circulating Tumor DNA
Keywords: Breast Cancer; Triple Negative Breast Cancer; Residual Cancer; Circulating Tumor DNA
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms; Neoplasm, Residual | interventions — atezolizumab; sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Atezolizumab and Sacituzumab govitecan (Experimental): Patients will receive the following treatment:
  Atezolizumab and Sacituzumab govitecan treatment will continue for 6 cycles (18 total weeks).
  * Atezolizumab intravenously (IV) at a pre-determined dose on day 1 in a 21-day cycle
  * Sacituzumab govitecan: intravenously (IV) at a pre-determined dose on days 1 and 8 in a 21-day cycle
  Interventions: Drug: Atezolizumab; Drug: Sacituzumab govitecan

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab is a type of antibody and is administered intravenously.
  Other Names: Tecentriq
Drug: Sacituzumab govitecan — Sacituzumab govitecan is an antibody drug conjugate and is administered intravenously
  Other Names: Trodelvy, IMMU-132

SUMMARY:
The purpose of this study is to determine if a combination of two drugs sacituzumab govitecan and atezolizumab works as a treatment for residual cancer in the breast or lymph nodes and have circulating tumor DNA in the blood.

This research study involves the following investigational drugs:

* Sacituzumab govitecan
* Atezolizumab

DETAILED DESCRIPTION:
This is an open label single-arm phase II study to evaluate the combination therapy of the antibody drug conjugate, sacituzumab govitecan, and the anti-PD-L1 antibody, atezolizumab, in patients with triple negative breast cancer.

The research study procedures include screening for eligibility and study treatment including laboratory evaluations, stool collection and follow up visits.

This research study involves the following investigational drugs:

* Sacituzumab govitecan
* Atezolizumab

Participants will receive study treatment for 18 weeks and will be followed for every 6 months for 3 years.

It is expected that about 40 people will take part in this research study.

This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug or drug combination works in treating a specific disease. "Investigational" means that the drug combination is being studied.

The U.S. Food and Drug Administration (FDA) has not approved atezolizumab (Tecentriq) for residual triple negative breast cancer but it has been approved for advanced triple negative breast cancer and other cancers. Atezolizumab is a protein that affects your immune system by blocking the PD-L1 pathway. The PD-L1 pathway controls your body's natural immune response, but for some types of cancer the immune system does not work as it should and is prevented from attacking tumors. Atezolizumab works by blocking the PD-L1 pathway, which may help your immune system identify and catch tumor cells.

The U.S. Food and Drug Administration (FDA) has not approved sacituzumab govitecan (Trodelvy) for your specific disease, but it has been approved for patients with metastatic triple-negative breast cancer who have been treated with 2 or more prior treatment regimens for their cancer. Sacituzumab govitecan is composed of a chemotherapy drug, called Irinotecan, which is attached to an antibody. Antibodies are proteins normally made by the immune system that bind to substances that don't belong in the body to prevent harm. The antibody in this study binds to certain types of cancer tumors.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed residual invasive breast cancer, in the breast and/or lymph node(s), following neoadjuvant chemotherapy. In the absence of residual invasive disease in the breast, lymph node must contain at least 2mm of invasive disease.
* HER2 negative in primary tumor pre-treatment by local pathology assessed according to current ASCO/CAP guidelines:

  * In situ hybridization non-amplified (ratio of HER2 to CEP17 < 2.0 or single probe average HER2 gene copy number < 4 signals/cell), OR
  * Immunohistochemistry (IHC) 0 or IHC 1+.
  * NOTE: If more than one test result is available and not all results meet the inclusion criterion definition, all results should be discussed with the Principal Investigator to establish eligibility
* ER and PR negative in primary tumor pre-treatment defined as < 10% of cells expressing hormonal receptors via IHC analysis by local laboratory assessment.
* Patients must have received neoadjuvant chemotherapy prior to breast surgery.
* Patients must be within 4 months of completion of all locoregional therapy (either last surgery or last dose of radiation, whichever is later) . Definitive breast surgery must have been performed and includes lumpectomy or mastectomy with pathologically clear margins (i.e. no ink on tumor). For patients undergoing lumpectomy, this must be followed by whole breast irradiation. Definitive surgery also includes axillary surgery, either sentinel lymph node biopsy or axillary lymph node dissection at the discretion of the attending surgeon.
* Evidence of ctDNA in blood sample collected after completion of all local and systemic neoadjuvant therapy (preoperative chemotherapy, surgery and radiation), confirmed by central testing. Detection of any tumor specific mutations (TSMs) within the sample will be considered positive for purposes of study eligibility.
* Concurrent receipt of bone modifying agents (bisphosphonates or rank-ligand inhibitors)is allowed.
* Prior treatment with an immune checkpoint inhibitor in the neoadjuvant setting is permitted.
* ECOG Performance Status of 0 or 1
* Men and women, age ≥ 18 years
* Adequate hematologic and organ function defined by the following:

  * ANC ≥ 1.5 × 109/L (1500/μL) without granulocyte colony-stimulating factor support
  * WBC count ≥ 2.5 × 109/L (2500/μL)
  * Absolute Lymphocyte count ≥ 0.5 × 109/L (500/μL)
  * Platelet count ≥ 100 × 109/L (100,000/μL)
  * Hemoglobin ≥ 90 g/L (9.0 g/dL), with or without transfusion
  * AST, ALT, and alkaline phosphatase (ALP) ≤ 2.5 × institutional upper limit of normal (ULN).
  * Serum bilirubin ≤ 1.5 × institutional ULN with the following exception:

    * Patients with known Gilbert syndrome: serum bilirubin level ≤ 3 × institutional ULN
  * Serum creatinine < 1.5 x institutional ULN
  * Creatinine clearance ≥30 mL/min as assessed by the Cockcroft-Gault equation
  * Serum albumin ≥ 25 g/L (2.5 g/dL)
  * For patients not receiving therapeutic anticoagulation: INR or aPTT ≤ 1.5 × institutional ULN
  * For patients receiving therapeutic anticoagulation: stable anticoagulant regimen
* Women of childbearing potential (pre-menopausal) must have a negative serum or urine pregnancy test within 7 days prior to start of therapy. A woman is defined as premenopausal if she is less than 12 months from last menstrual period with no identified cause other than menopause (medication induced amenorrhea is not acceptable). Pregnancy test is not required in women who are surgically sterile via bilateral salpingooophorectomy or hysterectomy.
* Women of childbearing potential and men must agree to use adequate contraception for the duration of protocol treatment and for 6 months after last dose of atezolizumab and 6 months after last dose of sacituzumab govitecan, whichever is later. Hormonal contraceptives are not acceptable (see section 5.6).
* Ability to understand and the willingness to sign a written informed consent document. Non-English speakers are eligible to participate but will be excluded from surveys/questionnaires unless the participant has a proxy available for translation.

Exclusion Criteria:

* Prior therapy with sacituzumab govitecan, irinotecan, or any topoisomerase I-containing antibody-drug conjugates at any time for early stage disease.
* Receipt of adjuvant chemotherapy (all chemotherapy prior to registration must have occurred in the preoperative setting)
* Prior hypersensitivity to atezolizumab or the excipients of atezolizumab or sacituzumab govitecan
* Clinical or radiographic evidence of metastatic disease
* Residual DCIS or LCIS alone without invasive cancer OR pT0N0i and pT0N1mic residual disease
* Concurrent enrollment on another investigational therapy trial
* Prior treatment-related toxicity must be resolved to ≤ Grade 1 prior to study enrollment with the exception of alopecia and peripheral neuropathy, prior to study enrollment.
* Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study
* Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
* Intercurrent illness including, but not limited to: ongoing or active infection requiring systemic therapy, active tuberculosis, serious liver disease such as cirrhosis, active bleeding diathesis, uncontrolled Type I or Type II diabetes mellitus, Grade ≥ 2 uncontrolled or untreated hypercholesterolemia, Hypertriglyceridemia or hypercalcemia
* Cardiovascular disease including: congestive heart failure of New York Heart Association Class III or IV, myocardial infarction (<6 months prior to enrollment) unstable angina pectoris, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease, in the opinion of the investigator
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Active (acute or chronic) autoimmune disease of any type except hypothyroidism on a thyroid-replacement hormone, celiac disease, or well-controlled psoriasis, eczema, lichen simplex chronicus or vitiligo.
* Impairment of gastrointestinal function or active gastrointestinal disease that may significantly alter the absorption of the study agents (e.g., ulcerative disease, uncontrolled nausea(> grade 2), vomiting (> grade 2), diarrhea (> grade 2), malabsorption syndrome or small bowel resection).
* Congenital long QT syndrome or screening QT interval corrected through use of Fridericia's formula >480 ms.
* Participants known to be positive for the human immunodeficiency virus (HIV), Hepatitis B antigen (HepBsAg), or Hepatitis C virus (HCV) RNA are ineligible.
* History of prior invasive breast cancer in either breast.
* Participants with history of prior malignancy other than breast cancer are eligible if they have been disease-free for at least 5 years prior to enrollment with the exception of patients with thyroid cancer that has been definitively treated without spread to regional lymph nodes.
* Treatment with strong strong UGT1A1 inhibitor or inducer within 4 weeks or 5 drug-elimination half-lives, whichever is longer, prior to initiation of study drug.
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine while on protocol treatment
* Known allergy or hypersensitivity to any of the study drugs or any of their excipients, including chimeric or humanized antibodies or fusion proteins and Chinese hamster ovary cell products or recombinant human antibodies
* Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor alpha agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during the course of the study, with the following exceptions:

  * Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible. o Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.
* Pregnant women are excluded from this study because the effects of sacituzumab govitecan and atezolizumab on a developing fetus are unknown. Breastfeeding should be discontinued prior to entry onto the study and for one month following the last dose of sacituzumab govitecan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-07-02 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of undetectable circulating tumor cfDNA- 6 Cycles | 18 Weeks
  Clearance of tumor cfDNA after 18 weeks, it will be tested using a one-sided one-sample binomial exact test (alpha 5%) against a null hypothesis value of 7% false negatives.

SECONDARY OUTCOMES:
Rate of undetectable circulating tumor cfDNA - 1 Cycle | 3 weeks
  Proportion of patients with undetectable circulating tumor cfDNA after 1 cycle of combination therapy
Rate of undetectable circulating tumor cfDNA - 3 Cycles | 9 weeks
  Proportion of patients with undetectable circulating tumor cfDNA after 3 cycles of combination therapy
Number of Participants With Treatment-Related Adverse Events | 18 Weeks
  Type, incidence and severity of adverse events (AEs) as graded by NCI CTCAE v5 criteria by 12 and 24 weeks.
Invasive disease-free survival (iDFS) Rate | 3 years
  Estimated disease-free survival (iDFS) Rate with 90% CI
Distant metastasis free survival (DMFS) Rate | 3 years
  Estimated metastasis free survival (DMFS) rate with 90% CI
Overall survival (OS) Rate | 3 years
  Estimate overall survival rate with 90% CI
3-year recurrence rate | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Mittendorf, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (7):
- United States (7):
  - University of California San Francisco, San Francisco, California
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center at Silver Cross Hospital, New Lenox, Illinois
  - University of Chicago Medical Center for Advanced Care Orland Park, Orland Park, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Pennsylvania-Abramson Cancer Center, Philadelphia, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Elizabeth Mittendorf, MD, PhD. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu